CLINICAL TRIAL: NCT01316419
Title: An Observational Study to Evaluate the Effects of Twynsta Tablets (Telmisartan and Amlodipine FDC, q.d.) With Life Style Modifications on Blood Pressure, Quality of Life, and Other Risk Factors in Korean Patients With Hypertension
Brief Title: Twynsta Study With Lifestyle Modifications in Korean Patients With Hypertension
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1235.42
Record Dates: First submitted 2011-03-15; First posted 2011-03-16 (Estimated); Results first posted 2015-07-27 (Estimated); Last update posted 2015-09-21 (Estimated); Status verified 2015-09

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Telmisartan; Amlodipine

STUDY DESIGN:
Time Perspective: Prospective

GROUPS / COHORTS (1):
- Patients with essential hypertension
  Interventions: Drug: Telmisartan; Drug: amlodipine

INTERVENTIONS:
Drug: Telmisartan — Telmisartan 40mg or 80mg
Drug: amlodipine — amlodipine 5mg or 10mg

SUMMARY:
This observational study is designed to evaluate the effects of Twynsta tablets with life style modifications on blood pressure, quality of life, and other risk factors in Korean patients with hypertension in a routine clinical practice setting.

DETAILED DESCRIPTION:
Study Design:

ELIGIBILITY:
Inclusion criteria:

1. Patients with essential hypertension whose blood pressure is not adequately controlled by amlodipine or telmisartan monotherapy (=140/90 mmHg, = 130/80 mmHg for those with diabetes or kidney disease)
2. Age = 19 years at enrollment
3. Male or female patient (or legally acceptable representative) willing and able to provide written informed consent

Exclusion criteria:

1. Patients with previous exposure to Twynsta
2. Patients with hypersensitivity to the active substances, or to dihydropyridine derivatives
3. Female patients at second and third trimesters of pregnancy
4. Female patients with lactation
5. Patients with biliary obstructive disorders
6. Patients with severe hepatic impairment
7. Patients with high grade aortic stenosis
8. Patients with shock
9. Patients with hereditary conditions such as intolerance with excipient of the products
10. Current participation in other clinical trials or observational studies

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Korean
Sampling Method: Probability Sample
Enrollment: 2089 (Actual)
Dates: Start 2011-03; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (55):
- South Korea (55):
  - Boehringer Ingelheim Investigational Site 15, Busan
  - Boehringer Ingelheim Investigational Site 37, Busan
  - Boehringer Ingelheim Investigational Site 42, Busan
  - Boehringer Ingelheim Investigational Site 55, Busan
  - Boehringer Ingelheim Investigational Site 54, Chonbuk
  - Boehringer Ingelheim Investigational Site 18, Chonnam
  - Boehringer Ingelheim Investigational Site 48, Chungcheong
  - Boehringer Ingelheim Investigational Site 46, Daegu
  - Boehringer Ingelheim Investigational Site 31, Daejeon
  - Boehringer Ingelheim Investigational Site 39, Daejeon
  - Boehringer Ingelheim Investigational Site 40, Daejeon
  - Boehringer Ingelheim Investigational Site 41, Daejeon
  - Boehringer Ingelheim Investigational Site 45, Daejeon
  - Boehringer Ingelheim Investigational Site 14, Deagu
  - Boehringer Ingelheim Investigational Site 25, Deagu
  - Boehringer Ingelheim Investigational Site 26, Deagu
  - Boehringer Ingelheim Investigational Site 44, Gangwon
  - Boehringer Ingelheim Investigational Site 24, Gwangju
  - Boehringer Ingelheim Investigational Site 32, Gwangju
  - Boehringer Ingelheim Investigational Site 11, Gyeonggi-do
  - Boehringer Ingelheim Investigational Site 13, Gyeonggi-do
  - Boehringer Ingelheim Investigational Site 16, Gyeonggi-do
  - Boehringer Ingelheim Investigational Site 21, Gyeonggi-do
  - Boehringer Ingelheim Investigational Site 23, Gyeonggi-do
  - Boehringer Ingelheim Investigational Site 30, Gyeonggi-do
  - Boehringer Ingelheim Investigational Site 43, Gyeonggi-do
  - Boehringer Ingelheim Investigational Site 47, Gyeonggi-do
  - Boehringer Ingelheim Investigational Site 5, Gyeonggi-do
  - Boehringer Ingelheim Investigational Site 6, Gyeonggi-do
  - Boehringer Ingelheim Investigational Site 9, Gyeonggi-do
  - Boehringer Ingelheim Investigational Site 35, Gyeongnam
  - Boehringer Ingelheim Investigational Site 51, Jeju City
  - Boehringer Ingelheim Investigational Site 52, Jeju City
  - Boehringer Ingelheim Investigational Site 17, Jungnam
  - Boehringer Ingelheim Investigational Site 19, Jungnam
  - Boehringer Ingelheim Investigational Site 8, Jungnam
  - Boehringer Ingelheim Investigational Site 12, Seoul
  - Boehringer Ingelheim Investigational Site 1, Seoul
  - Boehringer Ingelheim Investigational Site 20, Seoul
  - Boehringer Ingelheim Investigational Site 22, Seoul
  - Boehringer Ingelheim Investigational Site 27, Seoul
  - Boehringer Ingelheim Investigational Site 28, Seoul
  - Boehringer Ingelheim Investigational Site 29, Seoul
  - Boehringer Ingelheim Investigational Site 2, Seoul
  - Boehringer Ingelheim Investigational Site 33, Seoul
  - Boehringer Ingelheim Investigational Site 34, Seoul
  - Boehringer Ingelheim Investigational Site 36, Seoul
  - Boehringer Ingelheim Investigational Site 38, Seoul
  - Boehringer Ingelheim Investigational Site 3, Seoul
  - Boehringer Ingelheim Investigational Site 49, Seoul
  - Boehringer Ingelheim Investigational Site 4, Seoul
  - Boehringer Ingelheim Investigational Site 50, Seoul
  - Boehringer Ingelheim Investigational Site 53, Seoul
  - Boehringer Ingelheim Investigational Site 7, Seoul
  - Boehringer Ingelheim Investigational Site 10, Ulan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is an observational study to evaluate the effects of Twynsta tablets (Telmisartan and amlodipine fixed dose combination (FDC), once daily (q.d.)) with life style modifications on blood pressure, quality of life, and other risk factors in Korean patients with hypertension
Groups:
- Twynsta (Telmisartan and Amlodipine FDC) Tablets: Oral administration of Twynsta (Telmisartan and amlodipine FDC) tablets. The doses of telmisartan are 40 mg and 80 mg combined with either 5 mg or 10 mg of amlodipine. The dose combinations for telmisartan/amlodipine in the study are as follows: 40 mg/5 mg, 40 mg/10 mg and 80 mg/5 mg.
Period: Overall Study
Arm/Group | Twynsta (Telmisartan and Amlodipine FDC) Tablets
Started | 2089
Completed | 1824
Not Completed | 265
Not completed — Not treated | 103
Not completed — Violated inclusion/exclusion criterion | 143
Not completed — Lost to Follow-up | 19

BASELINE CHARACTERISTICS:
Population: All treated patients fulfilling the inclusion-exclusion criterias and who have completed the follow-up visits of the study.
Arm/Group | Twynsta (Telmisartan and Amlodipine FDC) Tablets
Number analyzed (Participants) | 1824
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.65 (13.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 778
  Male | 1046

OUTCOME MEASURES:

1. Primary Outcome: Mean Blood Pressure Change Systolic Blood Pressure (SBP) From Baseline After 24±2 Weeks of Treatment or at the Last Observation in Case of Early Withdrawal.
Description: The primary endpoint is the mean blood pressure change SBP from baseline after 24±2 weeks of treatment or at the last observation in case of early withdrawal.
  Baseline is defined as data collected on baseline visit.
Time Frame: baseline and 24±2 weeks
Population: All patients with a baseline and an endpoint blood pressure measurement.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Twynsta (Telmisartan and Amlodipine FDC) Tablets
Number analyzed (Participants) | 1662
mmHg | -21.81 (16.12)
Statistical Analysis 1: Comparison: Twynsta (Telmisartan and Amlodipine FDC) Tablets; Test type: Superiority or Other; p < 0.0001, Paired t test — Mean SBP change from baseline at the last visit will be analyzed by paired t-test

2. Secondary Outcome: Percentage of Patients Achieving Target Blood Pressure SBP/DBP <140/90 mmHg.
Description: Percentage of patients achieving target blood pressure SBP/DBP <140/90 mmHg is a key secondary endpoint.
Time Frame: 24±2 weeks
Population: All patients with a baseline and an endpoint blood pressure measurement.
Measure: Number; unit: percentage of participants
Arm/Group | Twynsta (Telmisartan and Amlodipine FDC) Tablets
Number analyzed (Participants) | 1662
percentage of participants | 74.07

3. Secondary Outcome: Percentage of Patients Achieving DBP Response
Description: Percentage of patients achieving DBP response (defined as mean seated DBP < 90 mmHg or a drop of ≥ 10 mmHg) is a key secondary endpoint.
Time Frame: 24±2 weeks
Population: All patients with a baseline and an endpoint blood pressure measurement.
Measure: Number; unit: percentage of participants
Arm/Group | Twynsta (Telmisartan and Amlodipine FDC) Tablets
Number analyzed (Participants) | 1662
percentage of participants | 88.99

4. Primary Outcome: Mean Blood Pressure Change Diastolic Blood Pressure (DBP) From Baseline After 24±2 Weeks of Treatment or at the Last Observation in Case of Early Withdrawal.
Description: The primary endpoint is the mean blood pressure change DBP from baseline after 24±2 weeks of treatment or at the last observation in case of early withdrawal.
  Baseline is defined as data collected on baseline visit.
Time Frame: baseline and 24±2 weeks
Population: All patients with a baseline and an endpoint blood pressure measurement.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Twynsta (Telmisartan and Amlodipine FDC) Tablets
Number analyzed (Participants) | 1662
mmHg | -13.48 (11.65)
Statistical Analysis 1: Comparison: Twynsta (Telmisartan and Amlodipine FDC) Tablets; Test type: Superiority or Other; p < 0.0001, Paired t test — Mean DBP change from baseline at the last visit will be analyzed by paired t-test

5. Secondary Outcome: Percentage of Patients Achieving SBP Response
Description: Percentage of patients achieving SBP response (defined as mean seated SBP < 140 mmHg or a drop of ≥ 10 mmHg) is a key secondary endpoint.
Time Frame: 24±2 weeks
Population: All patients with a baseline and an endpoint blood pressure measurement.
Measure: Number; unit: percentage of participants
Arm/Group | Twynsta (Telmisartan and Amlodipine FDC) Tablets
Number analyzed (Participants) | 1662
percentage of participants | 87.18

6. Secondary Outcome: Change From Baseline of Quality of Life Assessment Data Measured by World Health Organization Quality of Life (WHOQOL-BREF)- Physical Health Domain
Description: WHOQOL-BREF, an abbreviated 26 item version of the WHOQOL-100 was developed to enable a brief but accurate assessment of the quality of life.
  The Korean version of WHOQOL-BREF is valid and reliable in the assessment of quality of life in Koreans. The WHOQOL-BREF is based on the four domain structure (physical health, psychological, social relationships, and environment). It was designed to use 5-point scales for all questions (not at all, a little, moderately, mostly, and completely). The scale goes from 4 to 20 in each domain structure and 0 to 5 in overall score, a low value shows better physical health.
Time Frame: baseline and 24±2 weeks
Population: Patients with a baseline and an endpoint WHOQOL-BREF response
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Twynsta (Telmisartan and Amlodipine FDC) Tablets
Number analyzed (Participants) | 1490
scores on a scale | 0.07 (1.69)
Statistical Analysis 1: Comparison: Twynsta (Telmisartan and Amlodipine FDC) Tablets; Test type: Superiority or Other; p = 0.1099, Paired t test — The change of QOL data collected using the WHOQOL-BREF is analyzed by paired t-test

7. Secondary Outcome: Change From Baseline of Quality of Life Assessment Data Measured by World Health Organization Quality of Life (WHOQOL-BREF)- Psychological Domain
Description: as for outcome 6
Time Frame: baseline and 24±2 weeks
Population: All patients with a baseline and an endpoint blood pressure measurement.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Twynsta (Telmisartan and Amlodipine FDC) Tablets
Number analyzed (Participants) | 1490
scores on a scale | 0.11 (1.75)
Statistical Analysis 1: Comparison: Twynsta (Telmisartan and Amlodipine FDC) Tablets; Test type: Superiority or Other; p = 0.0197, Paired t test — The change of QOL data collected using the WHOQOL-BREF is analyzed by paired t-test

8. Secondary Outcome: Change From Baseline of Quality of Life Assessment Data Measured by World Health Organization Quality of Life (WHOQOL-BREF)- Social Relationships Domain
Description: as for outcome 6
Time Frame: baseline and 24±2 weeks
Population: Patients with a baseline and an endpoint WHOQOL-BREF response
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Twynsta (Telmisartan and Amlodipine FDC) Tablets
Number analyzed (Participants) | 1489
scores on a scale | -0.04 (2.31)
Statistical Analysis 1: Comparison: Twynsta (Telmisartan and Amlodipine FDC) Tablets; Test type: Superiority or Other; p = 0.4543, Paired t test — The change of QOL data collected using the WHOQOL-BREF is analyzed by paired t-test

9. Secondary Outcome: Change From Baseline of Quality of Life Assessment Data Measured by World Health Organization Quality of Life (WHOQOL-BREF)- Environment Domain
Description: as for outcome 6
Time Frame: baseline and 24±2 weeks
Population: Patients with a baseline and an endpoint WHOQOL-BREF response
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Twynsta (Telmisartan and Amlodipine FDC) Tablets
Number analyzed (Participants) | 1490
scores on a scale | 0.12 (1.97)
Statistical Analysis 1: Comparison: Twynsta (Telmisartan and Amlodipine FDC) Tablets; Test type: Superiority or Other; p = 0.0152, Paired t test — The change of QOL data collected using the WHOQOL-BREF is analyzed by paired t-test

10. Secondary Outcome: Change From Baseline of Quality of Life Assessment Data Measured by World Health Organization Quality of Life (WHOQOL-BREF)- Overall
Description: as for outcome 6
Time Frame: baseline and 24±2 weeks
Population: Patients with a baseline and an endpoint WHOQOL-BREF response
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Twynsta (Telmisartan and Amlodipine FDC) Tablets
Number analyzed (Participants) | 1490
scores on a scale | 0.03 (0.37)
Statistical Analysis 1: Comparison: Twynsta (Telmisartan and Amlodipine FDC) Tablets; Test type: Superiority or Other; p = 0.0013, Paired t test — The change of QOL data collected using the WHOQOL-BREF is analyzed by paired t-test

11. Secondary Outcome: EuroQol (EQ) Visual Analogue Scale (VAS)
Description: The EQ VAS records the respondent's self-rated health on a vertical, visual analogue scale where the endpoints are labelled 'best imaginable health state' and 'worst imaginable health state. The scale goes from 0 to 100, a low value shows better physical health.
Time Frame: baseline and 24±2 weeks
Population: Patients with a baseline and an endpoint EQ VAS response
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Twynsta (Telmisartan and Amlodipine FDC) Tablets
Number analyzed (Participants) | 1489
scores on a scale | 4.64 (16.24)
Statistical Analysis 1: Comparison: Twynsta (Telmisartan and Amlodipine FDC) Tablets; Test type: Superiority or Other; p < 0.0001, Paired t test — The change of QOL data collected using the EQ VAS is analyzed by paired t-test

12. Secondary Outcome: Percentage of Patients Achieving SBP/DBP < 130/80 mmHg Among Patients With Diabetes or Kidney Disease
Description: Percentage of patients achieving SBP/DBP < 130/80 mmHg among patients with diabetes or kidney disease
Time Frame: 24±2 weeks
Population: All patients with diabetes, kidney disease or both (diabetes + kidney disease)
Measure: Number; unit: percentage of participants
Arm/Group | Twynsta (Telmisartan and Amlodipine FDC) Tablets
Number analyzed (Participants) | 299
percentage of participants
  Diabetes (N=269) | 41.26
  Kidney Disease (N=20) | 40.00
  Diabetes + Kidney disease (N=10) | 50.00

13. Secondary Outcome: Mean Blood Lipid Change - Low Density Lipoprotein (LDL)-Cholesterol
Description: Mean blood lipid change from baseline - low density lipoprotein (LDL)-Cholesterol
Time Frame: baseline and 24±2 weeks
Population: Patients with medical history of hyperlipidemia and who have a baseline and an endpoint lipid profile measurement together with evaluation record on recommendations for lifestyle modifications.
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Twynsta (Telmisartan and Amlodipine FDC) Tablets
Number analyzed (Participants) | 124
mg/dl | -9.17 (29.16)
Statistical Analysis 1: Comparison: Twynsta (Telmisartan and Amlodipine FDC) Tablets; Test type: Superiority or Other; p = 0.0006, Paired t test — Mean LDL-C change from baseline at the last visit will be analyzed by paired t-test

14. Secondary Outcome: Mean Blood Lipid Change - High Density Lipoprotein (HDL)-Cholesterol
Description: Mean blood lipid change from baseline - high density lipoprotein (HDL)-Cholesterol
Time Frame: baseline and 24±2 weeks
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Twynsta (Telmisartan and Amlodipine FDC) Tablets
Number analyzed (Participants) | 134
mg/dl | 0.44 (6.34)
Statistical Analysis 1: Comparison: Twynsta (Telmisartan and Amlodipine FDC) Tablets; Test type: Superiority or Other; p = 0.4248, Paired t test — Mean HDL-C change from baseline at the last visit will be analyzed by paired t-test

15. Secondary Outcome: Mean Blood Lipid Change - Triglyceride
Description: Mean blood lipid change - Triglyceride
Time Frame: baseline and 24±2 weeks
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Twynsta (Telmisartan and Amlodipine FDC) Tablets
Number analyzed (Participants) | 134
mg/dl | -3.76 (74.12)
Statistical Analysis 1: Comparison: Twynsta (Telmisartan and Amlodipine FDC) Tablets; Test type: Superiority or Other; p = 0.5579, Paired t test — Mean Triglyceride change from baseline at the last visit will be analyzed by paired t-test

16. Secondary Outcome: Mean Blood Lipid Change - Total Cholesterol
Description: Mean blood lipid change - Total Cholesterol
Time Frame: baseline and 24±2 weeks
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Twynsta (Telmisartan and Amlodipine FDC) Tablets
Number analyzed (Participants) | 123
mg/dl | -9.62 (30.19)
Statistical Analysis 1: Comparison: Twynsta (Telmisartan and Amlodipine FDC) Tablets; Test type: Superiority or Other; p = 0.0006, Paired t-test — Mean total cholesterol change from baseline at the last visit will be analyzed by paired t-test

17. Secondary Outcome: Percentage of Patients Achieving Normal Body Mass Index (BMI)
Description: Percentage of patients achieving normal BMI (18.5 kg/sq.m to 24.9 kg/sq.m) are presented
Time Frame: 24±2 weeks
Population: Patients with a baseline and an endpoint BMI together with evaluation record on recommendations for lifestyle modifications.
Measure: Number; unit: percentage of participants
Arm/Group | Twynsta (Telmisartan and Amlodipine FDC) Tablets
Number analyzed (Participants) | 1392
percentage of participants | 45.62

18. Secondary Outcome: Percentage of Patients Who Complied With Each Category of Lifestyle Modification Recommendations at 12±2 Weeks
Description: Percentage of patients who complied with each category of lifestyle modification recommendations at 12±2 weeks
Time Frame: 12±2 weeks
Population: as for outcome 17
Measure: Number; unit: percentage of participants
Arm/Group | Twynsta (Telmisartan and Amlodipine FDC) Tablets
Number analyzed (Participants) | 1646
percentage of participants
  Physical activity | 71.87
  Well balanced diet | 84.33
  Dietary sodium reduction | 71.08
  Moderation of alcohol consumption | 82.38

19. Secondary Outcome: Percentage of Patients Who Complied With Each Category of Lifestyle Modification Recommendations at 24±2 Weeks
Description: Percentage of patients who complied with each category of lifestyle modification recommendations at 12±2 weeks
Time Frame: 24±2 weeks
Population: as for outcome 17
Measure: Number; unit: percentage of participants
Arm/Group | Twynsta (Telmisartan and Amlodipine FDC) Tablets
Number analyzed (Participants) | 1514
percentage of participants
  Physical activity | 77.21
  Well balanced diet | 87.38
  Dietary sodium reduction | 76.09
  Moderation of alcohol consumption | 83.49

20. Secondary Outcome: Incidence and Severity of Reported Adverse Events.
Description: Incidence as per the severity of reported adverse events is presented.
Time Frame: 24±2 weeks
Population: Patients having received at least one dose of Twynsta tablets
Measure: Number; unit: participants
Arm/Group | Twynsta (Telmisartan and Amlodipine FDC) Tablets
Number analyzed (Participants) | 1824
participants
  Mild | 220
  Moderate | 73
  Severe | 9

ADVERSE EVENTS:
Time Frame: All adverse events occurring during the course of the observational study (i.e., from signing the informed consent onwards through the observational phase); Up to 24±2 weeks
Arm/Group | Twynsta (Telmisartan and Amlodipine FDC) Tablets
Serious Adverse Events (participants affected / at risk) | 33/1824
Other Adverse Events (participants affected / at risk) | 0/1824
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Twynsta (Telmisartan and Amlodipine FDC) Tablets (N=1824)
Dizziness (Nervous system disorders) | 1
Cerebral infarction (Nervous system disorders) | 3
Cerebrovascular accident (Nervous system disorders) | 2
Vomiting (Gastrointestinal disorders) | 1
Pneumonia (Infections and infestations) | 2
Arthritis bacterial (Infections and infestations) | 1
Ophthalmic herpes zoster (Infections and infestations) | 1
Otitis media (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Asthenia (General disorders) | 1
Chest discomfort (General disorders) | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1
Fall (Injury, poisoning and procedural complications) | 2
Patella fracture (Injury, poisoning and procedural complications) | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1
Radius fracture (Injury, poisoning and procedural complications) | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1
Tibia fracture (Injury, poisoning and procedural complications) | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 1
Angina pectoris (Cardiac disorders) | 2
Coronary artery stenosis (Cardiac disorders) | 1
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Fibromatosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cataract (Eye disorders) | 1
Visual impairment (Eye disorders) | 1
Erectile dysfunction (Reproductive system and breast disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.